CLINICAL TRIAL: NCT03042364
Title: Cytokine Profile of the Uterine Secretome After Therapeutic Endometrial Scratching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Miacol-2017-3H
Record Dates: First submitted 2017-01-31; First posted 2017-02-03 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Infertility, Female
Keywords: Endometrium, Cytokines, Endometrial secretion, Implantation, Endometrial scratching
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (No Intervention): Standard treatment
- Intervention (Experimental): Endometrial scratching before standard treatment
  Interventions: Other: Pipelle de Cornier

INTERVENTIONS:
Other: Pipelle de Cornier — RCT with endometrial scratching prior to hormone treatment in ART. Aspiration of uterine secretion at transfer day
  Arms: Intervention

SUMMARY:
This study investigates the impact of endometrial scratching on endometrial secretion, when correlated to pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* IVF or ICSI patients with ≥1 previous implantation failure, despite transfer of a top quality embryo or blastocyst.
* Antagonist treatment
* FSH: 2-12 IU/L
* BMI: 18-32
* Regular menstrual cycle
* Written consent

Exclusion Criteria:

* Suspected intrauterine abnormalities Planned use of specialized media or AHA

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 150 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Cytokine profile of the uterine secretome after therapeutic endometrial scratching | Within 12 months
  The secretome is analyzed using a Multiplex analysis with 45 cytokines, chemokines and growth factors from ProcartaPlex Immunoassay Kit, Affymetrix, eBioscience. The samples are normalized for total protein content using a Nanodrop spectrophometer, and the protein composition is further determined by sodium dodecyl sulphate-polyacrylamide gel electropheresis (SDS-PAGE).
Immunoassay Kit: | Within 12 months
  BDNF, EGF, Eotaxin, FGF-2, GMCSF, GRO-alpha, HGF, IFN alpha, IFN gamma, IL-1RA, IL-1alpha, IL-1 beta, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12p70, IL-13, IL-15, IL17-A, IL-18, IL-21, IL-22, IL-23, IL-27, IL-31, IP-10, LIF, MCP-1, MIP-1 alpha, MIP-1 beta, NGF beta, RANTES, PDGF-BB, PÅIGF-1, SCF, SDF-1 alpha, TNF alpha, TNF beta, VEGF-A, VEGF-D

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (4):
  - Fertility Clinic,Aalborg University Hospital, Aalborg
  - Fertility Clinic, Herlev Hospital, Herlev
  - Fertility Clinic Horsens Hospital, Horsens
  - Fertility Clinic, Skive Hospital, Skive

IPD SHARING:
Plan to Share IPD: Undecided